CLINICAL TRIAL: NCT04532385
Title: Effect of a 12-week Administration of Green Tea Extract on Lipids in Patients With Type 2 Diabetes
Brief Title: Effect of Green Tea Extract on Lipids in Patients With Type 2 Diabetes
Acronym: HDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Profesor Investigador Titular A, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUCS-INTEC-MV-TEVE-002
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2; Dyslipidemias; Arterial Stiffness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Tea

STUDY DESIGN:
Intervention Model Description: patients were randomly assigned to receive green tea extract (sunphenon 90D, TAIYO international, Minneapolis, US) at a 400 mg/12 hrs dose or calcined magnesia (400 mg/12 hrs).
Who Masked: Participant, Investigator
Masking Description: An external pharmacy laboratory encapsulated the GTE and placebo, blinded and coded the study treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GTE (Experimental): Green tea extract, 400 mg every 12 hours for 12 weeks
  Interventions: Dietary Supplement: Green tea extract
- Placebo (Placebo Comparator): Calcined magnesia, 400 mg every 12 hours for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Green tea extract — 400 mg capsule
  Other Names: Sunphenon 90D
  Arms: GTE
Dietary Supplement: Placebo — 400 mg capsule
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
The main objectives of this study were to evaluate the effect of a 12-week supplementation with GTE (400 mg every 12 hours) on serum lipids, arterial stiffness and inflammatory cytokines in patients with T2DM.

DETAILED DESCRIPTION:
A 12 week randomized double-blind, placebo-controlled trial was conducted in patients with T2DM to evaluate the effect of green tea extract (sunphenon 90D, TAIYO international, Minneapolis, US) at a 400 mg/12 hrs dose or calcined magnesia (400 mg/12 hrs) on lipids, anthropometric variables, arterial stiffness and inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

- Patients with type 2 diabetes

Exclusion Criteria:

* Type 1 diabetes
* Smoking patients
* Ischemic heart disease
* Use of anti-inflammatory or antioxidant drugs
* Previously diagnosed liver or thyroid disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cholesterol at week 12 | baseline and week 12
  Measured using the Erba Manheim XL-100 automatic chemistry analyzer
Change from baseline in HDL at week 12 | baseline and week 12
  Measured using the Erba Manheim XL-100 automatic chemistry analyzer
Change from baseline in LDL at week 12 | baseline and week 12
  Calculated using Friedewald's equation for LDL (LDL = cholesterol - HDL - triglycerides/5)
Change from baseline in triglycerides at week 12 | baseline and week 12
  Measured using the Erba Manheim XL-100 automatic chemistry analyzer
Change from baseline in VLDL at week 12 | baseline and week 12
  Calculated using Friedewald's equation for VLDL (VLDL = triglycerides/5)
Change from baseline in augmentation index at week 12 | baseline and week 12
  Measured using the Omron HEM-9000AI tonometric system after resting in the sitting position for 5 minutes
Change from baseline in pulse pressure at week 12 | baseline and week 12
  Measured using the Omron HEM-9000AI tonometric system after resting in the sitting position for 5 minutes
Change from baseline in central systolic blood pressure at week 12 | baseline and week 12
  Measured using the Omron HEM-9000AI tonometric system after resting in the sitting position for 5 minutes
Change from baseline in IL-6 at week 12 | baseline and week 12
  Measurement was done using commercially available ELISA kits from Peprotech
Change from baseline in IL-1β at week 12 | baseline and week 12
  Measurement was done using commercially available ELISA kits from Peprotech
Change from baseline in TNF-α at week 12 | baseline and week 12
  Measurement was done using commercially available ELISA kits from Peprotech

SECONDARY OUTCOMES:
Change from baseline in glucose at week 12 | baseline and week 12
  Measured using the Erba Manheim XL-100 automatic chemistry analyzer
Change from baseline in Hemoglobin A1c at week 12 | baseline and week 12
  Measured using the Bio-Rad Variant Classic Hemoglobin testing system
Change from baseline in systolic blood pressure at week 12 | baseline and week 12
  Measured using the Omron HEM-9000AI tonometric system after resting in the sitting position for 5 minutes
Change from baseline in diastolic blood pressure at week 12 | baseline and week 12
  Measured using the Omron HEM-9000AI tonometric system after resting in the sitting position for 5 minutes
Change from baseline in IMC at week 12 | baseline and week 12
  Measured with the Tanita TBF-215 Body Composition Analyzer
Change from baseline in body fat percentage at week 12 | baseline and week 12
  Measured with the Tanita TBF-215 Body Composition Analyzer
Change from baseline in fat mass at week 12 | baseline and week 12
  Measured with the Tanita TBF-215 Body Composition Analyzer
Change from baseline in lean mass at week 12 | baseline and week 12
  Measured with the Tanita TBF-215 Body Composition Analyzer
Change from baseline in body water at week 12 | baseline and week 12
  Measured with the Tanita TBF-215 Body Composition Analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Gavish B, Izzo JL Jr. Arterial Stiffness: Going a Step Beyond. Am J Hypertens. 2016 Nov 1;29(11):1223-1233. doi: 10.1093/ajh/hpw061. PMID 27405964
- [Background] Shirwany NA, Zou MH. Arterial stiffness: a brief review. Acta Pharmacol Sin. 2010 Oct;31(10):1267-76. doi: 10.1038/aps.2010.123. Epub 2010 Aug 30. PMID 20802505
- [Background] Lessiani G, Santilli F, Boccatonda A, Iodice P, Liani R, Tripaldi R, Saggini R, Davi G. Arterial stiffness and sedentary lifestyle: Role of oxidative stress. Vascul Pharmacol. 2016 Apr;79:1-5. doi: 10.1016/j.vph.2015.05.017. Epub 2015 Jun 2. PMID 26044182
- [Background] Virdis A, Taddei S. Endothelial Dysfunction in Resistance Arteries of Hypertensive Humans: Old and New Conspirators. J Cardiovasc Pharmacol. 2016 Jun;67(6):451-7. doi: 10.1097/FJC.0000000000000362. PMID 26808712
- [Background] de Maat MP, Pijl H, Kluft C, Princen HM. Consumption of black and green tea had no effect on inflammation, haemostasis and endothelial markers in smoking healthy individuals. Eur J Clin Nutr. 2000 Oct;54(10):757-63. doi: 10.1038/sj.ejcn.1601084. PMID 11083483
- [Background] Stokes GS, Barin ES, Gilfillan KL. Effects of isosorbide mononitrate and AII inhibition on pulse wave reflection in hypertension. Hypertension. 2003 Feb;41(2):297-301. doi: 10.1161/01.hyp.0000049622.07021.4f. PMID 12574098
- [Background] Vlachopoulos C, Terentes-Printzios D, Ioakeimidis N, Rokkas K, Samentzas A, Aggelis A, Kardara D, Stefanadis C. Beneficial effect of vardenafil on aortic stiffness and wave reflections. J Clin Pharmacol. 2012 Aug;52(8):1215-21. doi: 10.1177/0091270011413586. Epub 2011 Sep 27. PMID 21953573
- [Background] Jeyaseelan L, Rao PS. Methods of determining sample sizes in clinical trials. Indian Pediatr. 1989 Feb;26(2):115-21. PMID 2753525
- [Background] Liu CY, Huang CJ, Huang LH, Chen IJ, Chiu JP, Hsu CH. Effects of green tea extract on insulin resistance and glucagon-like peptide 1 in patients with type 2 diabetes and lipid abnormalities: a randomized, double-blinded, and placebo-controlled trial. PLoS One. 2014 Mar 10;9(3):e91163. doi: 10.1371/journal.pone.0091163. eCollection 2014. PMID 24614112
- [Background] Kohara K, Tabara Y, Oshiumi A, Miyawaki Y, Kobayashi T, Miki T. Radial augmentation index: a useful and easily obtainable parameter for vascular aging. Am J Hypertens. 2005 Jan;18(1 Pt 2):11S-14S. doi: 10.1016/j.amjhyper.2004.10.010. PMID 15683726
- [Background] Cui R, Yamagishi K, Muraki I, Hayama-Terada M, Umesawa M, Imano H, Li Y, Eshak ES, Ohira T, Kiyama M, Okada T, Kitamura A, Tanigawa T, Iso H; CIRCS investigators. Association between markers of arterial stiffness and atrial fibrillation in the Circulatory Risk in Communities Study (CIRCS). Atherosclerosis. 2017 Aug;263:244-248. doi: 10.1016/j.atherosclerosis.2017.06.918. Epub 2017 Jun 22. PMID 28683363
- [Background] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736
- [Background] Quezada-Fernandez P, Trujillo-Quiros J, Pascoe-Gonzalez S, Trujillo-Rangel WA, Cardona-Muller D, Ramos-Becerra CG, Barocio-Pantoja M, Rodriguez-de la Cerda M, Nerida Sanchez-Rodriguez E, Cardona-Munoz EG, Garcia-Benavides L, Grover-Paez F. Effect of green tea extract on arterial stiffness, lipid profile and sRAGE in patients with type 2 diabetes mellitus: a randomised, double-blind, placebo-controlled trial. Int J Food Sci Nutr. 2019 Dec;70(8):977-985. doi: 10.1080/09637486.2019.1589430. Epub 2019 May 14. PMID 31084381
- [Background] Brown AL, Lane J, Coverly J, Stocks J, Jackson S, Stephen A, Bluck L, Coward A, Hendrickx H. Effects of dietary supplementation with the green tea polyphenol epigallocatechin-3-gallate on insulin resistance and associated metabolic risk factors: randomized controlled trial. Br J Nutr. 2009 Mar;101(6):886-94. doi: 10.1017/S0007114508047727. Epub 2008 Aug 19. PMID 18710606
- [Background] Onakpoya I, Spencer E, Heneghan C, Thompson M. The effect of green tea on blood pressure and lipid profile: a systematic review and meta-analysis of randomized clinical trials. Nutr Metab Cardiovasc Dis. 2014 Aug;24(8):823-36. doi: 10.1016/j.numecd.2014.01.016. Epub 2014 Jan 31. PMID 24675010
- [Background] Marinovic MP, Morandi AC, Otton R. Green tea catechins alone or in combination alter functional parameters of human neutrophils via suppressing the activation of TLR-4/NFkappaB p65 signal pathway. Toxicol In Vitro. 2015 Oct;29(7):1766-78. doi: 10.1016/j.tiv.2015.07.014. Epub 2015 Jul 15. PMID 26187476
- [Background] Bogdanski P, Suliburska J, Szulinska M, Stepien M, Pupek-Musialik D, Jablecka A. Green tea extract reduces blood pressure, inflammatory biomarkers, and oxidative stress and improves parameters associated with insulin resistance in obese, hypertensive patients. Nutr Res. 2012 Jun;32(6):421-7. doi: 10.1016/j.nutres.2012.05.007. Epub 2012 Jun 20. PMID 22749178
- [Background] Cox AJ, West NP, Cripps AW. Obesity, inflammation, and the gut microbiota. Lancet Diabetes Endocrinol. 2015 Mar;3(3):207-15. doi: 10.1016/S2213-8587(14)70134-2. Epub 2014 Jul 22. PMID 25066177